CLINICAL TRIAL: NCT01326091
Title: Operative Patient Positioning in Lumbar Fusion Surgery and Its Impact on Spinal Sagittal Balance and Surgeon Satisfaction
Brief Title: Patient Positioning in Lumbar Fusion Surgery and Its Impact on Spinal Sagittal Balance and Surgeon Satisfaction
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient study support
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00028159
Record Dates: First submitted 2011-03-29; First posted 2011-03-30 (Estimated); Last update posted 2015-06-23 (Estimated); Status verified 2015-05

CONDITIONS: Intervertebral Disk Degeneration
Keywords: Lumbar fusion surgery
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Positioning (No Intervention)
- Hyperlordotic Positioning (Active Comparator): Hyperlordotic positioning will be achieved through pelvic pads positioned low on iliac crest to maximize lumbar hyperlordosis and increased hip flexion with as many pillows as tolerated at thighs and knees to allow for increased sacral slope. Regular position will involve the pelvic pads at above or iliac crest and without extra pillows at thighs and legs.
  Interventions: Other: Hyperlordotic Positioning

INTERVENTIONS:
Other: Hyperlordotic Positioning — Hyperlordotic positioning will be achieved through pelvic pads positioned low on iliac crest to maximize lumbar hyperlordosis and increased hip flexion with as many pillows as tolerated at thighs and knees to allow for increased sacral slope. Regular position will involve the pelvic pads at above or iliac crest and without extra pillows at thighs and legs.
  Arms: Hyperlordotic Positioning

SUMMARY:
This is a parallel, randomized controlled trial comparing two types of patient positioning and their effect on radiologic measures (pre-surgery visit, in the operating room prior to surgery, at the conclusion of surgery, and at 3 weeks after surgery at patients' postoperative visits) as well as surgeon satisfaction (prior to the end of the surgery) and patient outcomes using patient self reported scales (pre-surgery, post surgery at 3 weeks follow-up).

DETAILED DESCRIPTION:
The investigators are evaluating how patient positioning affects radiologic metrics as well as surgeon satisfaction (surgeon being blinded to positioning). Patients will be allocated to either a hyperlordotic or a standard positioning group by computer generated randomization. Surgeons will perform all of their standard techniques to promote lordosis with instrumentation. Adult patients, ages 18-65, undergoing lumbar surgical fusion will be asked to participate.

ELIGIBILITY:
Inclusion Criteria:

* Adults patients, aged between 18 and 65 years of age
* Patients undergoing lumbar fusion for degenerative conditions

Exclusion Criteria:

* Patients < 18 years of age or > 65 years of age
* Patients who have a history of metastatic disease
* Patients who currently have a pending workman's compensation claim
* Patients who have had a previous spinal surgery
* Patients who have or have had a spinal infection
* Patients who have a spinal deformity, such as scoliosis
* Women who are pregnant
* Inpatients

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2011-03; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
To assess if the specific intra-operative positioning affects post-operative sagittal alignment | Will be assessed during immediate post-operative period (day 1) as well as 3 weeks post-operatively
  X-rays will be performed at patients' pre-surgery visit, in the operating room prior to surgery and at the conclusion of surgery, and at 3 weeks after surgery at patients' postoperative visit. The specifics of the pelvic parameters will be measured at these visits. Also, the patient will complete VAS, ODI (Davidson, 2002; Fairbank, 2000 ), and WHOQOL-BREF prior to surgery and at 3 weeks follow-up. We will collect data on any complications occurring in the perioperative period till 3 weeks after surgery

SECONDARY OUTCOMES:
Surgeon satisfaction with operative patient positioning | During surgery (day 1)
  Satisfaction ratings with regard to comfort in performing decompression and fusion will be collected by the coordinator prior to the end of the surgery to ensure that the surgeon remains blinded to allocation. It will be measured through a questionnaire using a series of verbal analog scales where 0 is completely unsatisfied and 10 is completely satisfied, the surgeon's degree of satisfaction with patient positioning and ease or difficulty in performing the surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Oren N Gottfried, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States